CLINICAL TRIAL: NCT01397786
Title: A Long-term, Phase 3, Multicenter, Open-label Trial to Evaluate the Safety and Tolerability of Oral OPC-34712 as Maintenance Treatment in Adults With Schizophrenia
Brief Title: Safety and Tolerability Study of Oral OPC-34712 as Maintenance Treatment in Adults With Schizophrenia
Acronym: ZENITH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-10-237
Record Dates: First submitted 2011-07-11; First posted 2011-07-20 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-34712 (Experimental)
  Interventions: Drug: OPC-34712

INTERVENTIONS:
Drug: OPC-34712 — Phase A: 1-2 mgs/day by mouth, max of 4 wks.
  Phase B: 1-4 mgs/day by mouth, up to 52 weeks

SUMMARY:
The purpose of this study is to assess the long-term safety, tolerability and efficacy of oral OPC-34712 as monotherapy in adults with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severely debilitating mental illness that affects approximately 1% of the world population. Hallucinations and delusions are the most striking characteristic positive symptoms of schizophrenia; however, more subtle negative symptoms (eg, social withdrawal and lack of emotion, energy, and motivation) may also be present. The first antipsychotics developed for the treatment of schizophrenia were effective against positive symptoms, but showed little efficacy for negative symptoms and were also associated with a high incidence of side effects. Second generation antipsychotics, represent a significant advancement in the treatment of psychotic disorders because they are effective and at the same time exhibit fewer side effects than first generation antipsychotics. Although generally safer than first generation antipsychotics, the second-generation antipsychotics are not devoid of undesirable side effects such as Hyperprolactinemia and weight gain. In addition, the safety of these drugs vary considerably.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 65 years of age, with a diagnosis of schizophrenia, as defined by DSM-IV-TR criteria
2. Outpatient status at last visit of Trial 331-10-230 or Trial 331-10-231
3. Willing to discontinue all prohibitive psychotropic medications to meet protocol required washouts prior to and during the trial period.
4. Other protocol specific inclusion criteria may apply.

Exclusion Criteria:

1. Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving study drug
2. Subjects with a current DSM-IV-TR Axis I diagnosis of:

   * Schizoaffective disorder
   * MDD
   * Bipolar disorder
   * Delirium, dementia, amnestic or other cognitive disorder
   * Borderline, paranoid, histrionic, schizotypal, schizoid or antisocial personality disorder
3. Subjects presenting with a first episode of schizophrenia
4. Other protocol specific exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Skuban, M.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (127):
- United States (49):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Springdale, Arkansas
  - Anaheim, California
  - Cerritos, California
  - Escondido, California
  - Garden Grove, California
  - Glendale, California
  - Long Beach, California
  - National City, California
  - Oakland, California
  - Oceanside, California
  - Pico Rivera, California
  - San Diego, California
  - Torrance, California
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Leesburg, Florida
  - Maitland, Florida
  - Miami, Florida
  - Miami Springs, Florida
  - North Miami, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Joliet, Illinois
  - Oak Brook, Illinois
  - Overland Park, Kansas
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Flowood, Mississippi
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Buffalo, New York
  - Cedarhurst, New York
  - Jamaica, New York
  - Rochester, New York
  - Staten Island, New York
  - Dayton, Ohio
  - Allentown, Pennsylvania
  - Norristown, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Richmond, Virginia
  - Kirkland, Washington
- Canada (2):
  - Burlington, Ontario
  - Chatham, Ontario
- Colombia (4):
  - Barranquilla
  - Bello
  - Bogotá
  - Pereira
- Croatia (2):
  - Rijeka
  - Zagreb
- Japan (4):
  - Fujisawa-shi, Kanagawa
  - Kumamoto, Kumamoto
  - Kunigami-gun, Okinawa
  - Sakai-shi, Osaka
- Latvia (5):
  - Daugavpils
  - Jelgava
  - Liepāja
  - Riga
  - Strenči
- Malaysia (6):
  - Kota Bharu, Kelantan
  - Kuala Lumpur, Kuala Lumpur
  - Kajang, Selangor
  - Ipoh
  - Jalan Greentown
  - Sabak Bernam
- Mexico (3):
  - Col. Florida, Mexico City
  - Monterrey, Nuevo León
  - San Luis Potosí City, San Luis Potos
- Philippines (3):
  - Cebu City
  - Davao City
  - Manila
- Poland (3):
  - Choroszcz
  - Gdansk
  - Lodz
- San Juan, Puerto Rico
- Romania (9):
  - Arad
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Focşani
  - Iași
  - Piteşti
  - Târgovişte
- Russia (10):
  - Arkhangelsk
  - Moscow
  - Moscow Region
  - Nizhny Novgorod
  - Petrozavodsk
  - Saint Petersburg
  - Samara
  - Saratov
  - Tomsk
  - Village Nikolskoe
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Novi Kneževac
  - Novi Sad
- Slovakia (4):
  - Bratislava
  - Michalovce
  - Rimavská Sobota
  - Rožňava
- South Korea (2):
  - Incheon
  - Seoul
- Taiwan (4):
  - Kashsiung
  - New Taipei City
  - Taipei
  - Taoyuan
- Turkey (Türkiye) (2):
  - Diyarbakır
  - Kocaeli
- Ukraine (10):
  - Chernihiv
  - Dnipropetrovsk
  - Hlevakha
  - Kharkiv
  - Kherson, Vil. Stepanivka
  - Kyiv
  - Lviv
  - Odesa
  - Simferopol
  - Vinnytsia

REFERENCES:
- [Derived] Correll CU, He Y, Therrien F, MacKenzie E, Meehan SR, Weiss C, Hefting N, Hobart M. Effects of Brexpiprazole on Functioning in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. J Clin Psychiatry. 2022 Mar 1;83(2):20m13793. doi: 10.4088/JCP.20m13793. PMID 35235720
- [Derived] Marder SR, Meehan SR, Weiss C, Chen D, Hobart M, Hefting N. Effects of Brexpiprazole Across Symptom Domains in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. Schizophr Bull Open. 2021 May 1;2(1):sgab014. doi: 10.1093/schizbullopen/sgab014. eCollection 2021 Jan. PMID 34901863
- [Derived] Newcomer JW, Eriksson H, Zhang P, Weiller E, Weiss C. Changes in metabolic parameters and body weight in brexpiprazole-treated patients with acute schizophrenia: pooled analyses of phase 3 clinical studies. Curr Med Res Opin. 2018 Dec;34(12):2197-2205. doi: 10.1080/03007995.2018.1498779. Epub 2018 Jul 27. PMID 29985680
- [Derived] Forbes A, Hobart M, Ouyang J, Shi L, Pfister S, Hakala M. A Long-Term, Open-Label Study to Evaluate the Safety and Tolerability of Brexpiprazole as Maintenance Treatment in Adults with Schizophrenia. Int J Neuropsychopharmacol. 2018 May 1;21(5):433-441. doi: 10.1093/ijnp/pyy002. PMID 29415258
- [Derived] Kane JM, Skuban A, Hobart M, Ouyang J, Weiller E, Weiss C, Correll CU. Overview of short- and long-term tolerability and safety of brexpiprazole in patients with schizophrenia. Schizophr Res. 2016 Jul;174(1-3):93-98. doi: 10.1016/j.schres.2016.04.013. Epub 2016 May 14. PMID 27188270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in a total of 1072 participants (1044 of whom entered the open-label treatment phase) at 202 trial sites in the following 18 countries: Japan, Korea, Malaysia, Philippines, Taiwan, Croatia, Latvia, Poland, Romania, Russia, Serbia, Turkey, Ukraine, Columbia, Mexico, Canada, Puerto Rico, and United States of America (USA).
Pre-assignment Details: Enrollment was drawn from eligible participants who could potentially benefit from monotherapy treatment with oral brexpiprazole for schizophrenia and included rollover participants from the double-blind, phase-3 efficacy trials (ie, Trial NCT01393613, Trial NCT01396421, and Trial NCT01668797) and de novo participants from select sites.
Groups:
- Prior Brexpiprazole: Participants who rolled over from, and received blinded brexpiprazole in, one of the randomized, double-blind, placebo-controlled Phase 3 efficacy studies (Vector, NCT01396421; Beacon, NCT01393613; and Equator, NCT01668797); all received 1-4 mg of daily treatment with open label brexpiprazole in trial NCT01397786 .
- Prior Placebo: Participants who rolled over from, and received blinded placebo in, one of the randomized, double-blind, placebo-controlled Phase 3 efficacy studies (Vector, NCT01396421; Beacon, NCT01393613; and Equator, NCT01668797); all received 1-4 mg of daily treatment with open label brexpiprazole in trial NCT01397786.
- De Novo: Participants who had not previously participated in a brexpiprazole clinical study and who received 1-4 mg of daily treatment with open label brexpiprazole in trial NCT01397786.
Period: Phase A
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo
Started | 12 (Subjects in NCT01668797 Phase A at IA-related study termination rolled over to NCT01397786 Phase A.) | 0 | 227
Completed | 12 | 0 | 199
Not Completed | 0 | 0 | 28
Not completed — Lost to Follow-up | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 8
Not completed — Subject Met Withdrawal Criteria | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 5
Not completed — Lack of Efficacy | 0 | 0 | 1
Period: Phase B
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo
Started | 611 | 204 | 229
Completed | 308 | 109 | 91
Not Completed | 303 | 95 | 138
Not completed — Lost to Follow-up | 22 | 12 | 22
Not completed — Adverse Event | 109 | 23 | 27
Not completed — Subject Met Withdrawal Criteria | 38 | 5 | 38
Not completed — Physician Decision | 9 | 1 | 3
Not completed — Withdrawal by Subject | 102 | 45 | 30
Not completed — Protocol Deviation | 1 | 2 | 4
Not completed — Lack of Efficacy | 22 | 7 | 14

BASELINE CHARACTERISTICS:
Groups:
- Prior Brexpiprazole: Participants who rolled over from, and received blinded brexpiprazole in, one of the randomized, double-blind, placebo-controlled Phase 3 efficacy studies (Vector, NCT01396421; Beacon, NCT01393613; and Equator, NCT01668797); all received 1-4 mg of daily treatment with open label brexpiprazole in trial NCT01397786.
- Total: Total of all reporting groups
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 611 | 204 | 257 | 1072
Age, Continuous [Mean (Standard Deviation); unit: participants] | 38.5 (10.8) | 39.6 (10.8) | 44.1 (11.1) | 40.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 79 | 85 | 409
  Male | 366 | 125 | 172 | 663

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: A treatment-emergent adverse event (TEAE) is defined as an AE that started after start of investigational medicinal product (IMP) treatment; or if the event was continuous from baseline and was serious, IMP-related, or resulted in death, discontinuation, interruption or reduction of IMP.
Time Frame: From Baseline up to 52 Weeks
Population: Safety sample included those participants who had at least one post-baseline efficacy evaluation for Positive and Negative Syndrome Scale (PANSS) total score.
Measure: Number; unit: percentage of participants
Groups:
- Total: Participants who rolled over from, and received blinded brexpiprazole/placebo in, one of the randomized, double blind, placebo controlled Phase 3 efficacy studies (Vector, NCT01396421;Beacon, NCT01393613; and Equator, NCT01668797); or de novo patients, All received 1-4 mg of daily treatment with open label brexpiprazole in trial NCT01397786.
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 605 | 202 | 224 | 1031
percentage of participants
  With AEs | 60.2 | 56.4 | 65.2 | 60.5
  With TEAEs | 60.0 | 56.4 | 65.2 | 60.4
  With SAEs | 14.9 | 8.9 | 11.2 | 12.9

2. Secondary Outcome: Mean Change From Baseline in Positive and Negative Syndrome Scale Total Score
Description: The PANSS consisted of 3 subscales with 30 symptom constructs (positive subscale (7): delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/perseckion, and hostility; negative subscale (7): blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and conversation flow, stereotyped thinking and general psychopathology subscale (16): somatic concern, anxiety, guilt feelings, tension, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgment and insight, disturbance of volition, poor impulse control, preoccupation, and active social avoidance). Severity was rated on 7-point scale with scores 1 (absence) & 7 (extremely severe). The PANSS total score was sum of rating scores for 7 positive, 7 negative, and 16 general psychopathology subscale items of PANSS panel.
Time Frame: From Baseline up to 52 Weeks
Population: The Efficacy Sample included participants in the Safety Sample who had at least 1 post-baseline efficacy evaluation for PANSS Total Score.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 223 | 1012
Units on a scale
  At Week 26 (Participant count=375,134,123,632) | -6.90 (12.90) | -12.50 (14.90) | -6.60 (13.60) | -8.00 (13.60)
  At Week 52 (Participant count= 226,93,91,410) | -11.0 (14.40) | -18.40 (16.90) | -8.80 (12.60) | -12.20 (15.00)
  At Last Visit (Participant count=591,198,223,1012) | -3.80 (16.70) | -9.70 (18.70) | -3.50 (14.30) | -4.90 (16.80)

3. Secondary Outcome: Mean Change From Baseline in PANSS Positive Subscale Score
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. In positive subscale, the 7 positive symptom constructs were: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility.
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 123 | 1012
Units on a scale
  At Week 26 (Participant count=375,134,123,632) | -2.10 (4.50) | -4.10 (5.40) | -1.70 (4.30) | -2.40 (4.70)
  At Week 52 (Participant count=226,93,91,410) | -3.20 (4.60) | -5.80 (5.20) | -2.30 (4.10) | -3.60 (4.80)
  At Last Visit (Participant count=591,198,223,1012) | -0.90 (5.90) | -2.80 (6.40) | -1.00 (4.90) | -1.30 (5.80)

4. Secondary Outcome: Mean Change From Baseline in PANSS Negative Subscale Score
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. In negative subscale the severity was rated for the following 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking.
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 223 | 1012
Units on a scale
  At Week 26 (Participant count=375,134,123,632) | -1.40 (3.70) | -2.40 (4.30) | -1.30 (3.80) | -1.60 (3.90)
  At Week 52 (Participant count=226,93,91,410) | -2.70 (4.50) | -3.70 (5.40) | -2.00 (3.70) | -2.80 (4.60)
  At Last Visit (Participant count=591,198,223,1012) | -1.00 (4.10) | -2.40 (5.00) | -0.60 (4.20) | -1.20 (4.30)

5. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression - Severity of Illness Scale Score
Description: The severity of illness for each participant was rated using the CGI-S. To perform this assessment, the investigator were to answer the following question: "Considering your total clinical experience with this particular population, how mentally ill was the participant at that time?" Response choices include: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 223 | 1012
Units on a scale
  At at Week 26 (Participant count=375,134,123,632) | -0.35 (0.79) | -0.60 (0.98) | -0.24 (0.88) | -0.38 (0.86)
  At Week 52 (Participant count=226,93,91,410) | -0.55 (0.86) | -0.97 (0.98) | -0.48 (0.86) | -0.63 (0.91)
  At Last Visit (Participant count=591,198,223,1012) | -0.14 (1.04) | -0.46 (1.12) | -0.17 (0.88) | -0.21 (1.03)

6. Secondary Outcome: Mean Change From Baseline in Personal and Social Performance Scale Total Score
Description: The PSP was a validated clinician-rated scale that measured personal and social functioning in four domains: socially useful activities (e.g, work and study), personal and social relationships, self-care, and disturbing and aggressive behaviors. Impairment in each of these domains was rated as absent, mild, manifest, marked, severe, or very severe. These ratings were then converted to a total score based on a 100-point scale using algorithms to identify the appropriate 10-point interval, and the rater's judgment that determined the total score within the 10-point interval. Participants with a PSP total score of 71 to 100 were considered to have mild functional difficulty. Scores of 31 to 70 represented manifest disabilities of various degrees and ratings of 1 to 30 indicated minimal functioning that required intense support and/or supervision.
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 123 | 1012
Units on a scale
  At Week 26 (Participant count=366,134,123,623) | 4.50 (9.70) | 6.50 (11.30) | 4.50 (9.00) | 4.90 (10.00)
  At Week 52 (Participant count=223,93,91,407) | 7.00 (10.60) | 9.60 (11.90) | 7.60 (10.80) | 7.70 (11.00)
  At Last Visit (Participant count=569,196,219,984) | 1.80 (12.40) | 5.10 (12.80) | 2.70 (11.00) | 2.70 (12.20)

7. Secondary Outcome: Mean Clinical Global Impression - Improvement Score
Description: The efficacy of study medication was rated for each participant using the CGI-I. The investigator rated the participant's total improvement whether or not it was due to the drug treatment. All responses were compared to the participant's condition at Screening/Baseline (i.e, Week 6 visit of Protocol NCT00905307). Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 598 | 198 | 123 | 1012
Units on a scale
  At Week 26 (Participant count=381,134,123,638) | 3.00 (1.13) | 2.77 (0.99) | 3.00 (1.13) | 2.95 (1.10)
  At Week 52 (Participant count=226,93,91,410) | 2.66 (1.13) | 2.26 (0.97) | 2.76 (1.09) | 2.59 (1.10)
  At Last Visit (Participant count=598,198,223,1019) | 3.31 (1.43) | 2.96 (1.33) | 3.30 (1.27) | 3.24 (1.38)

8. Secondary Outcome: Response Rate
Description: Response rate was defined as a reduction of ≥ 30% from Baseline in PANSS total score or CGI-I score of 1 (very much improved) or 2 (much improved) at the Last Visit.
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 605 | 202 | 224 | 1031
percentage of participants | 34.2 | 42.6 | 27.2 | 34.3

9. Secondary Outcome: Discontinuation Rate for Lack of Efficacy
Description: Discontinuation rate for the participants who discontinued due to lack of efficacy were examined.
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 605 | 202 | 224 | 1031
percentage of participants | 3.6 | 3.5 | 6.3 | 4.2

10. Secondary Outcome: Mean Change From Baseline in Positive and Negative Syndrome Scale Excited Component Score
Description: The PEC score consisted of five PANSS items: excitement (P4), hostility (P7), tension (G4), uncooperativeness (G8), and poor impulse control (G14). Each of the items were rated on a scale of 1 (absent) to 7 (extreme). The PEC scores ranged from 5 (not present) to 35 (extremely severe).
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 123 | 1012
Units on a scale
  At Week 26 (Participant count=375,134,123,632) | -0.60 (3.10) | -1.80 (3.70) | -0.70 (3.10) | -0.90 (3.30)
  At Week 52 (Participant count=226,93,91,410) | -1.20 (3.20) | -2.60 (3.40) | -1.00 (2.90) | -1.50 (3.20)
  At Last Visit (Participant count=591,198,223,1012) | 0.10 (4.10) | -0.90 (4.20) | -0.30 (3.50) | -0.20 (4.00)

11. Secondary Outcome: Mean Change From Baseline in PANSS Marder Factor Scores - Positive Symptoms Score
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The positive factor score was the sum of the 8 components (delusions (P1), hallucinatory behavior (P3), grandiosity (P5), suspiciousness/persecution (P6), stereotyped thinking (N7), somatic concern (G1), unusual thought content (G9) and lack of judgment and insight (G12)) of the positive symptoms scale (range: 8 - best possible outcome to 56 - worst possible outcome).
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Prior Placebo; De Novo: Participants who rolled over from, and received blinded brexpiprazole in, one of the randomized, double-blind, placebo-controlled Phase 3 efficacy studies (Vector, NCT01396421; Beacon, NCT01393613; and Equator, NCT01668797); all received 1-4 mg of daily treatment with open label brexpiprazole in trial NCT01397786.
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 123 | 1012
Units on a scale
  At Week 26 (Participant count=375,134,123,632) | -2.60 (4.80) | -4.70 (5.50) | -2.00 (5.20) | -2.90 (5.10)
  At Week 52 (Participant count=226,93,91,410) | -3.90 (5.20) | -6.60 (5.70) | -2.60 (4.80) | -4.20 (5.40)
  At Last Visit (Participant count=591,198,223,1012) | -1.60 (5.90) | -3.50 (6.50) | -1.30 (5.00) | -1.90 (5.90)

12. Secondary Outcome: Mean Change From Baseline in PANSS Marder Factor Scores - Negative Symptoms Score
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The negative factor score is the sum of the 7 items (blunted affect (N1), emotional withdrawal (N2), poor rapport (N3), passive/apathetic social withdrawal (N4), lack of spontaneity and conversation flow (N6), motor retardation (G7) and active social avoidance (G16)) of the negative subscale (range: 8 - best possible outcome to 56 - worst possible outcome).
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 123 | 1012
Units on a scale
  At Week 26 (Participant count=375,134,123,632) | -1.50 (3.60) | -2.20 (4.00) | -1.70 (4.10) | -1.70 (3.80)
  At Week 52 (Participant count=226,93,91,410) | -2.60 (4.30) | -3.90 (5.00) | -2.20 (3.80) | -2.80 (4.40)
  At Last Visit (Participant count=591,198,223,1012) | -1.00 (4.10) | -2.30 (5.10) | -0.70 (4.10) | -1.20 (4.40)

13. Secondary Outcome: Mean Change From Baseline in PANSS Marder Factor Scores - Disorganized Thought Score
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The disorganized thoughts factor score is the sum of score from the 7 items (conceptual disorganization (P2), difficulty in abstract thinking (N5), mannerisms and posturing (G5), disorientation (G10), poor attention (G11), disturbance of volition (G13) and preoccupation (G15)) on the disorganized thoughts subscale (range: 7 - best possible outcome to 49 - worst possible outcome).
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 123 | 1012
Units on a scale
  At Week 26 (Participant count=375,134,123,632) | -1.70 (3.30) | -2.60 (3.50) | -1.70 (3.50) | -1.90 (3.40)
  At Week 52 (Participant count=226,93,91,410) | -2.90 (3.70) | -3.70 (4.60) | -2.30 (3.70) | -2.90 (4.00)
  At Last Visit (Participant count=591,198,223,1012) | -1.20 (4.20) | -2.20 (4.50) | -0.90 (4.00) | -1.40 (4.20)

14. Secondary Outcome: Mean Change From Baseline in PANSS Marder Factor Scores - Hostility/ Excitement Score
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The uncontrolled hostility/excitement factor score is the sum of score from the 4 items (excitement (P4), hostility (P7), uncooperativeness (G8) and poor impulse control (G14)) on the uncontrolled hostility/excitement subscale (range: 4 - best possible outcome to 28 - worst possible outcome).
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 123 | 1012
Units on a scale
  At Week 26 (Participant count=375,134,123,632) | -0.40 (2.70) | -1.40 (3.10) | -0.60 (2.60) | -0.60 (2.80)
  At Week 52 (Participant count=226,93,91,410) | -0.80 (2.70) | -1.90 (2.90) | -0.90 (2.30) | -1.10 (2.70)
  At Last Visit (Participant count=591,198,223,1012) | 0.20 (3.40) | -0.70 (3.50) | -0.30 (3.00) | -0.10 (3.40)

15. Secondary Outcome: Mean Change From Baseline in PANSS Marder Factor Scores - Anxiety/Depression Score
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The anxiety/depression factor score is the sum of score from the 4 items (anxiety (G2), guilt feelings (G3), tension (G4) and depression (G6)) on the anxiety/depression subscale (range: 4 - best possible outcome to 28 - worst possible outcome).
Time Frame: From Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | De Novo | Total
Number analyzed (Participants) | 591 | 198 | 123 | 1012
Units on a scale
  At Week 26 (Participant count=375,134,123,632) | -0.70 (2.60) | -1.50 (3.00) | -0.70 (3.40) | -0.90 (2.90)
  At Week 52 (Participant count=226,93,91,410) | -0.90 (2.50) | -2.40 (2.90) | -0.80 (3.50) | -1.20 (2.90)
  At Last Visit (Participant count=591,198,223,1012) | -0.20 (3.20) | -0.90 (3.40) | -0.40 (3.80) | -0.40 (3.40)

ADVERSE EVENTS:
Time Frame: The trial required that participants be actively monitored for AEs up to 30 (+2) days after the last dose of study drug, up to 52 weeks.
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with use of a drug in humans, whether or not considered drug related. Serious adverse event (SAE) includes any AE that meets the either one or more seriousness criteria mentioned in the study protocol. An immediately Reportable Event (IRE) was defined as any SAE, AE/pregnancy cases that necessitates discontinuation of IMP/potential Hy's Law cases. Included participants who received at least 1 dose of open-label IMP.
Groups:
- De Novo (Phase A): Participants underwent cross-titration to oral brexpiprazole for 4 weeks in Phase A. DeNovo participants in Phase A received brexpiprazole monotherapy starting dose of 2 mg daily at the conversion Week 4 visit (baseline visit of Phase B). Participants who received at least 1 dose of study drug were included in this phase.
  NOTE: 12 participants from the trial P33110232 were excluded in this analysis.
- Prior Brexpiprazole (Phase B): Participants who rolled over from, and received blinded brexpiprazole in, one of the randomized, double-blind, placebo-controlled Phase 3 efficacy studies (Vector, NCT01396421; Beacon, NCT01393613; and Equator, NCT01668797); all received 1-4 mg of daily treatment with open label brexpiprazole in trial NCT01397786. Participants who received at least 1 dose of study drug were included in this phase.
  NOTE: Six participants from the trial P33110231 were excluded in this analysis.
- Prior Placebo (Phase B): Participants who rolled over from, and received blinded placebo in, one of the randomized, double-blind, placebo-controlled Phase 3 efficacy studies (Vector, NCT01396421; Beacon, NCT01393613; and Equator, NCT01668797); all received 1-4 mg of daily treatment with open label brexpiprazole in trial NCT01397786.
  Participants who received at least 1 dose of study drug were included in this phase.
  NOTE: One participant each from the trials P33110230 and P33110231 were excluded in this analysis.
- De Novo (Phase B): Participants who had not previously participated in a brexpiprazole clinical study and who received 1-4 mg of daily treatment with open label brexpiprazole in trial NCT01397786. Participants who received at least 1 dose of study drug were included in this phase.
  NOTE: Five participants from Phase B - Denovo were excluded in this analysis.
Arm/Group | De Novo (Phase A) | Prior Brexpiprazole (Phase B) | Prior Placebo (Phase B) | De Novo (Phase B)
Serious Adverse Events (participants affected / at risk) | 4/226 | 90/605 | 18/202 | 25/224
Other Adverse Events (participants affected / at risk) | 0/226 | 166/605 | 53/202 | 95/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo (Phase A) (N=226) | Prior Brexpiprazole (Phase B) (N=605) | Prior Placebo (Phase B) (N=202) | De Novo (Phase B) (N=224)
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 2 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 2 | 68 | 12 | 10
Psychotic disorder (Psychiatric disorders) | 1 | 7 | 3 | 4
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2
Schizophrenia, Paranoid type (Psychiatric disorders) | 0 | 1 | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo (Phase A) (N=226) | Prior Brexpiprazole (Phase B) (N=605) | Prior Placebo (Phase B) (N=202) | De Novo (Phase B) (N=256)
Weight increased (Investigations) | 0 | 47 | 15 | 23
Akathisia (Nervous system disorders) | 0 | 22 | 14 | 14
Headache (Nervous system disorders) | 0 | 42 | 14 | 24
Agitation (Psychiatric disorders) | 0 | 30 | 7 | 23
Insomnia (Psychiatric disorders) | 0 | 51 | 17 | 32
Hypertension (Vascular disorders) | 0 | 10 | 2 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.